CLINICAL TRIAL: NCT00491868
Title: Switch and Maintenance Study of Intravenous Injections of R744 to Hemodialysis Patients ( Phase III, Double Blind Study in Comparison With Epoetin Beta).
Brief Title: Clinical Study of R744 to Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JH20876
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Hemodialysis Patients
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: R744; Drug: rHuEPO placebo
- 2 (Experimental)
  Interventions: Drug: R744; Drug: rHuEPO placebo
- 3 (Active Comparator)
  Interventions: Drug: rHuEPO; Drug: R744 placebo
- 4 (Active Comparator)
  Interventions: Drug: rHuEPO; Drug: R744 placebo

INTERVENTIONS:
Drug: R744 — 100μg/4week for 8 weeks, then 50~250μg/4week for 16 weeks
  Other Names: methoxy polyethylene glycol-epoetin beta
  Arms: 1
Drug: R744 — 150μg/4week for 8 weeks, then 50~250μg/4week for 16 weeks
  Other Names: methoxy polyethylene glycol-epoetin beta
  Arms: 2
Drug: rHuEPO — 2250IU or 3000IU(i.v.) 2 or 3 times/week for 8 weeks, then 750~9000IU(i.v.)/1~3week for 16 weeks
  Arms: 3
Drug: rHuEPO — 4500IU or 6000IU(i.v.) 2 or 3times/week for 8 weeks, then 750~9000IU(i.v.)/1~3week for 16 weeks
  Arms: 4
Drug: R744 placebo — 0 μg/4week for 24 weeks
  Arms: 3; 4
Drug: rHuEPO placebo — 0 IU 2 or 3 times/week for 8 weeks, then 1~3 times/week for 16 weeks
  Arms: 1; 2

SUMMARY:
This study used as the comparative drug (epoetin beta) will assess the efficacy and safety of intravenous injections of R744 in renal anemia patients on Hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been receiving hemodialysis 3 times a week for at least 12 weeks before registration
* Patients aged ≥ 20 years at the time of obtaining consent
* Patients who have been receiving a rHuEPO preparation at least once a week for at least 8 weeks before registration
* Within 4 weeks before registration, patients who have been receiving a rHuEPO preparation 750IU (3 times a week), 1,500IU (twice a week (1st and 2nd hemodialysis day of the week, or1st and 3rd hemodialysis day of the week)), 1,500IU (3 times a week), or 3,000IU (twice a week (1st and 2nd hemodialysis day of the week, or1st and 3rd hemodialysis day of the week)), and patients who have not change dosage and administration.
* Patients whose pre-dialysis Hb concentrations has been between ≥ 9.0 g/dL and ≤12.0 g/dL and mean value of pre-dialysis Hb concentrations has been between ≥ 9.5 g/dL and ≤11.5 g/dL determined at the beginning of each week within 8 weeks before registration
* Patients whose transferrin saturation has been ≥ 20 % or ferritin has been ≥ 100ng/mL at any time point within 8 weeks before registration

Exclusion Criteria:

* Patients with hardly controllable hypertension (patients whose diastolic blood pressure has been ≥ 100 mmHg on more than 1/3 of the determining occasions within 12 weeks before registration)
* Patients with congestive cardiac failure (≥ Class III in NYHA cardiac function classification)
* Female patients who are pregnant, lactating, possibly pregnant or not willing to take a contraceptive measure in the period from the day of starting the treatment with the study drug to 90 days after the day of the last dose of the study drug
* Patients with complication of myocardial infarction, pulmonary infarction or cerebral infarction (excluding asymptomatic cerebral infarction)
* Patients confirmed to have serious allergy or serious drug allergy (shock, anaphylactoid symptom)
* Patients hypersensitive to a rHuEPO preparation
* Patients with malignant tumor (including hemic malignant tumor), severe infection, systemic hemic disease (osteomyelodysplasia syndrome, hemoglobinopathy, etc.), hemolytic anemia or apparent hemorrhagic lesion such as digestive tract hemorrhage
* Patients who have received an anabolic hormone preparation, testosterone enanthate, testosterone propionate, methyltestosterone or mepitiostane within 12 weeks before registration
* Patients who have received another investigational drug within 12 weeks before registration
* Patients who have received R744 before registration
* Patients whose AST(GOT) value ≥ 100 IU/L or ALT(GPT) value ≥ 100 IU/L before registration
* Patients who have received erythrocyte transfusion within 16 weeks before registration
* Patients for whom a surgical operation accompanied by marked bleeding is planned during the study period
* In addition, patients who are judged as ineligible to participate in this study by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Variation of Hb concentration from baseline Hb concentration in evaluation period | week 17~24

SECONDARY OUTCOMES:
Rate of patients who maintain Hb concentration in the range of baseline ± 1.0g/dL and maintain Hb concentration in the range of ≥ 9.0g/dL and ≤ 12.0g/dL in evaluation period | week 17~24
Rate of patients who maintain Hb concentration within ±1.0g/dL of reference Hb | week 17~24
Adverse events | throughout study
Laboratory measurements | throughout study
Vital signs, standard 12-lead ECG | throughout study
Anti-R744 antibody titer | throughout study
Anti-Epoetin beta antibody titer | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Takanori Baba, Study Chair — Chugai Pharmaceutical,Clinical Research Department 2
Locations (5):
- Japan (5):
  - Chugoku/Shikoku region, Chugoku/Shikoku
  - Chubu region, Chūbu
  - Kanto/Koshinetsu region, Kanto/Koshinetsu
  - Kinki/Hokuriku region, Kinki/Hokuriku
  - Kyusyu region, Kyusyu